CLINICAL TRIAL: NCT00892021
Title: An Ascending Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NSA-789 Administered Orally to Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: Study Evaluating the Effects of Multiple Doses of NSA-789 in Subjects With Schizophrenia or Schizoaffective Disorder
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 3230A1-1003
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2009-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSA-789 (Experimental): Active study drug
  Interventions: Drug: NSA-789
- Placebo (Placebo Comparator): Inactive study drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NSA-789
  Arms: NSA-789
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety of multiple doses of NSA-789 in subjects with schizophrenia or schizoaffective disorder. This study will also assess how NSA-789 is absorbed and eliminated, and its effect, if any, on the brain.

ELIGIBILITY:
Inclusion:

* Men or women of non childbearing potential (WONCBP) aged 18 to 50 years, inclusive.
* Currently under the care of a physician for psychiatric illness.
* Clinical diagnosis of schizophrenia or schizo affective disorder in the opinion of the study psychiatrist based on review of all available clinical data.

Exclusion:

* Any unstable medical or psychiatric condition, which may prevent the successful and safe completion of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by adverse events, monitoring of safety variables (ECGs, vital signs, laboratory test results) | 6 months

SECONDARY OUTCOMES:
Tolerability as measured through the reporting of adverse events; Pharmacokinetic as measured by the concentrations of NSA-789 in blood; Pharmacodynamics as measured by the results of psychiatric ratings and neurologic evaluations. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Rockville, Maryland, United States